CLINICAL TRIAL: NCT02286089
Title: Phase I/IIa Dose Escalation Safety and Efficacy Study of Human Embryonic Stem Cell-Derived Retinal Pigment Epithelium Cells Transplanted Subretinally in Patients With Advanced Dry-Form Age-Related Macular Degeneration (Geographic Atrophy)
Brief Title: Safety and Efficacy Study of OpRegen for Treatment of Advanced Dry-Form Age-Related Macular Degeneration
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GR44172; NCT06674993 (obsolete NCT alias)
Record Dates: First submitted 2014-11-02; First posted 2014-11-07 (Estimated); Results first posted 2023-03-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OpRegen (Experimental): Up to 12 legally blind subjects with best corrected visual acuity of 20/200 or less in first three cohorts and 12 subjects with best corrected visual acuity of 20/64 and 20/250 in fourth cohort
  Interventions: Biological: OpRegen

INTERVENTIONS:
Biological: OpRegen — Targeted dose of 50,000 - 200,000 cells will be delivered into the subretinal space.

SUMMARY:
The main objective of the study is evaluation of the safety and tolerability of OpRegen - Human embryonic stem cell-derived retinal pigment epithelial (RPE) cells. The study will also include initial exploration of the ability of transplanted OpRegen cells to engraft, survive, and moderate disease progression.

DETAILED DESCRIPTION:
OpRegen® is a cell-based product composed of retinal pigment epithelial (RPE) cells, derived from human embryonic stem cells (hESC) and administered as a cell suspension either in ophthalmic Balanced Salt Solution Plus (BSS Plus) or in CryoStor® 5 (Thaw-and-Inject, TAI). This is a Phase I/IIa, dose-escalation, evaluating safety and tolerability of OpRegen transplantation to patients with progressive dry-AMD. The study includes also initial exploration of efficacy.

A total of approximately 24 subjects will be enrolled. The subjects should be 50 years of age and older, with non-neovascular (dry) AMD, who have funduscopic findings of GA in the macula, with absence of additional concomitant ocular disorders. The subjects will be divided into four cohorts, according to their best corrected visual acuity (BCVA) and administered OpRegen dose.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and older;
* Diagnosis of dry (non-neovascular) age related macular degeneration in both eyes;
* Funduscopic findings of dry age-related macular degeneration (AMD) with progressive geographic atrophy in the macula;
* Best corrected central visual acuity equal or less than 20/200 in cohorts 1-3 and 20/64-20/250 in cohort 4 in the study eye by ETDRS vision testing;
* Vision in the non-operated eye must be better than or equal to that in the operated eye;
* Subjects with sufficiently good health to allow participation in all study-related procedures and complete the study follow up period (based on medical records);
* Ability to undergo a vitreoretinal surgical procedure under monitored anesthesia care;
* Blood counts, blood chemistry, coagulation and urinalysis without abnormal significance;
* Negative for tuberculosis (TB) (cohort 4), human immunodeficiency virus (HIV), hepatitis B (HBC), and hepatitis C virus (HCV), negative for cytomegalovirus (CMV) Immunoglobulin (IgM) and Epstein-Barr Virus (EBV) IgM or asymptomatic in the opinion of the investigator (cohort 4);
* No history of malignancy (other than a non-melanoma skin cancer). For cancers in remission for more then 5 years enrollment is allowed with concurred documented approval of principal investigator and oncologist prior to enrollment;
* Willing to defer all future blood and tissue donation;
* Able to understand study procedures and willing to sign informed consent.

Exclusion Criteria:

* Evidence of neovascular AMD by history, as well as by clinical exam, fluorescein angiography (FA), or ocular coherence tomography (OCT) at baseline in either eye;
* History or presence of diabetic retinopathy, vascular occlusions, uveitis, Coat's disease, uncontrolled glaucoma, cataract or media opacity preventing posterior pole visualization or any significant ocular disease other than AMD that has compromised or could compromise vision in the study eye and confound analysis of the primary outcome;
* History of retinal detachment repair in the study eye;
* Axial myopia greater than -6 diopters;
* At least 2 months following cataract removal in the study eye and Yttrium Aluminum Garnet (YAG) laser capsulotomy in the study eye in the past 4 weeks and any other ocular surgery in the study eye in the past 3 months prior to implantation;
* History of cognitive impairments or dementia;
* Contraindication for systemic immunosuppression;
* History of any condition other than AMD associated with choroidal neovascularization in the study eye (e.g. pathologic myopia or presumed ocular histoplasmosis);
* Any type of systemic disease or its treatment, in the opinion of the Investigator, including any medical condition (controlled or uncontrolled) that could be expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical status of the participant to a significant degree or put the patient at special risk.
* Pregnancy or breastfeeding;
* Current participation in another clinical study. Past participation (within 6 months) in any clinical study of a drug administered systemically or to the eye.
* Currently receiving aspirin, aspirin containing products and/or any other coagulation modifying drugs which cannot be discontinued 7 days prior to surgery;
* History of cancer (other than a non-melanoma skin cancer). For cancers in remission more than five years ago, enrollment is allowed with concurred documented approval of principal investigator and oncologist prior to enrollment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2031-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- United States (3):
  - West Coast Retina Medical Group, San Francisco, California
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
- Israel (4):
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Aweidah H, Matsevich C, Khaner H, Idelson M, Ejzenberg A, Reubinoff B, Banin E, Obolensky A. Survival of Neural Progenitors Derived from Human Embryonic Stem Cells Following Subretinal Transplantation in Rodents. J Ocul Pharmacol Ther. 2023 Jun;39(5):347-358. doi: 10.1089/jop.2022.0161. Epub 2023 May 4. PMID 37140896

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment into the study was staggered with 4 week intervals between the first 3 cohorts to allow for data safety monitory board (DSMB) review. Accumulated data of participants was reviewed by the DSMB before continuation to Cohort 4. All four cohorts were then followed in parallel.
Groups:
- Cohort 1: Participants in cohort 1 with Best Corrected Visual Acuity (BCVA) of 20/200 or less received a single subretinal delivery of the low dose of OpRegen on Day 0.
- Cohort 2: Participants in cohort 2 with BCVA of 20/200 or less received a single subretinal delivery of the high dose of OpRegen on Day 0.
- Cohort 3: Additional participants in cohort 3 with BCVA of 20/200 or less received a single subretinal delivery of the high dose of OpRegen on Day 0.
- Cohort 4: Participants in cohort 4 with BCVA of 20/64 to 20/250 received a single subretinal delivery of the high dose of OpRegen on Day 0.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 3 | 3 | 6 | 12
Completed | 2 | 2 | 0 | 0
Not Completed | 1 | 1 | 6 | 12
Not completed — Ongoing in Study | 1 | 1 | 4 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.4 (2.7) | 74.4 (8.7) | 80.4 (9.9) | 78.1 (8.2) | 76.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 6 | 13
  Male | 1 | 0 | 4 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 6 | 12 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. The AE's were graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 3.0.
Time Frame: From study start till 12 months following last subject dosed, plus up to 90 days (up to approximately 6.5 years)
Population: Safety Population included all participants who received OpRegen in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 6 | 12
percentage of participants
  Blood and lymphatic system disorders | 33.3 | 33.3 | 0 | 8.3
  Cardiac disorders | 33.3 | 0 | 0 | 8.3
  Ear and labyrinth disorders | 66.7 | 33.3 | 16.7 | 8.3
  Endocrine disorders | 0 | 0 | 0 | 8.3
  Eye disorders | 100 | 100 | 100 | 100
  Gastrointestinal disorders | 66.7 | 66.7 | 0 | 33.3
  General disorders and administration site conditions | 66.7 | 100 | 50.0 | 16.7
  Infections and infestations | 100 | 66.7 | 50.0 | 33.3
  Injury, poisoning and procedural complications | 66.7 | 100 | 50.0 | 16.7
  Investigations | 100 | 66.7 | 33.3 | 75.0
  Metabolism and nutrition disorders | 0 | 0 | 16.7 | 33.3
  Musculoskeletal and connective tissue disorders | 66.7 | 66.7 | 0 | 33.3
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 0 | 33.3 | 50.0 | 25.0
  Nervous system disorders | 0 | 33.3 | 50.0 | 33.3
  Psychiatric disorders | 0 | 0 | 0 | 8.3
  Surgical and medical procedures | 100 | 66.7 | 0 | 16.7
  Skin and subcutaneous tissue disorders | 33.3 | 33.3 | 33.3 | 8.3
  Vascular disorders | 0 | 0 | 16.7 | 16.7
  Product issues | 66.7 | 0 | 0 | 0
  Renal and urinary disorders | 0 | 0 | 33.3 | 0
  Respiratory, thoracic and mediastinal disorders | 66.7 | 66.7 | 16.7 | 0

2. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP)
Time Frame: Baseline, Month 12
Population: Safety Population included all participants who received OpRegen in the study.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 6 | 12
mmHg
  Baseline | 13.3 (2.3) | 14.0 (0.0) | 13.7 (3.7) | 14.6 (3.1)
  Change from Baseline at Month 12: number analyzed (Participants) | 3 | 3 | 5 | 12
  Change from Baseline at Month 12 | 1.0 (2.6) | 1.0 (1.7) | -0.4 (2.5) | -0.6 (1.4)

3. Secondary Outcome: Change From Baseline in Geographic Atrophy (GA) Lesion Area
Description: The GA lesion area was based on available Fundus Autofluorescence (FAF) imaging data by a central reading center.
Time Frame: Baseline, Month 12
Population: Efficacy Population included all participants who received OpRegen in the study and for whom imaging data were available.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 6 | 12
mm^2
  Baseline | 13.5 (6.4) | 18.5 (10.6) | 9.4 (2.0) | 7.4 (2.9)
  Change from Baseline at Month 12: number analyzed (Participants) | 2 | 1 | 3 | 11
  Change from Baseline at Month 12 | 2.3 (1.9) | 1.6 (NA) — NA: Standard deviation cannot be calculated for 1 participant. | 2.5 (4.0) | 1.8 (0.8)

4. Secondary Outcome: Change From Baseline in Visual Acuity
Description: Change from baseline in visual acuity was measured by retro illuminated ETDRS chart from 4 meters distance. Visual acuity was reported as the number of letters read correctly.
Time Frame: Baseline, Month 12
Population: Efficacy Population included all participants who received OpRegen in the study.
Measure: Mean (Standard Deviation); unit: number of letters
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 6 | 12
number of letters
  Baseline | 20.0 (18.0) | 14.3 (7.2) | 29.8 (6.8) | 44.8 (7.5)
  Change from Baseline at Month 12: number analyzed (Participants) | 3 | 3 | 5 | 12
  Change from Baseline at Month 12 | 15.7 (34.2) | 3.0 (8.7) | -1.4 (17.8) | 7.6 (8.7)

5. Secondary Outcome: Change From Baseline in National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) Quality of Life
Description: The NEI VFQ-25 is a 25 item patient-reported questionnaire. The composite score ranges from 0-100 with the higher score indicating better visual function.
Time Frame: Baseline, Month 12
Population: Efficacy Population included all participants who received OpRegen in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 6 | 12
score on a scale
  Baseline | 50.3 (15.3) | 42.9 (6.0) | 46.9 (18.8) | 62.2 (13.8)
  Change from Baseline at Month 12: number analyzed (Participants) | 3 | 3 | 5 | 11
  Change from Baseline at Month 12 | 5.1 (10.8) | -5.7 (17.6) | 3.1 (18.2) | 3.7 (11.4)

ADVERSE EVENTS:
Time Frame: From study start till 12 months following last subject dosed, plus up to 90 days (up to approximately 6.5 years)
Description: Safety Population included all participants who received OpRegen in the study.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 2/6 | 4/12
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=6) | Cohort 4 (N=12)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=6) | Cohort 4 (N=12)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conductive deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 2 (2) | 4 (6) | 1 (1)
Macular fibrosis (Eye disorders) | 2 (2) | 3 (6) | 5 (7) | 6 (9)
Subretinal fluid (Eye disorders) | 2 (6) | 2 (2) | 1 (2) | 2 (3)
Age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anterior chamber disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 3 (3) | 3 (3) | 8 (9)
Conjunctival hyperaemia (Eye disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Conjunctival irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Eyelid haematoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyphaema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic atrophy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Punctate keratitis (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Retinal cyst (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal depigmentation (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 5 (5)
Retinal pigmentation (Eye disorders) | 2 (3) | 3 (5) | 2 (6) | 2 (2)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retinopathy proliferative (Eye disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Retinoschisis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Implant site atrophy (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer helicobacter (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ocular procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Angiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
B-lymphocyte count abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood immunoglobulin G increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
CD4/CD8 ratio decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Free prostate-specific antigen increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wound healing normal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tunnel vision (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract discomfort (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Cataract operation (Surgical and medical procedures) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Dental implantation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intra-ocular injection (Surgical and medical procedures) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Posterior lens capsulotomy (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blebitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Conjunctival bleb (Eye disorders) | 0 (0) | 0 (0) | 0/5 (0) | 1 (1)
Corneal disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cystoid macular oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Detachment of retinal pigment epithelium (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 5 (5)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Iritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pinguecula (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pouchitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine renal clearance increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immunosuppressant drug level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SGOT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vital dye staining cornea present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subconjunctival injection procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anterior Chamber inflammation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT02286089/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT02286089/SAP_001.pdf